CLINICAL TRIAL: NCT01639573
Title: Campath-1h as Immunoablative Therapy for Children and Adolescents With Treatment Refractory Systemic Sclerosis
Brief Title: Campath-1h Phase I/II Pilot Trial as Immunoablative Therapy for Refractory Systemic Sclerosis
Acronym: CAMPATH-1H
Status: Withdrawn | Type: Observational
Why Stopped: The study has stopped due to no patient enrollment unable to meet the study criteria
Sponsor: Children's Hospital Los Angeles (Other)
Responsible Party: Principal Investigator, Diane Brown, Co-Principal Investigator, Children's Hospital Los Angeles
Other Study IDs: CCI-11-00077
Record Dates: First submitted 2012-06-18; First posted 2012-07-12 (Estimated); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Scleroderma
Keywords: Patients with Scleroderma
MeSH Terms: conditions — Scleroderma, Diffuse | interventions — Alemtuzumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Campath — Pediatric patients with dcSSc are eligible for the clinical trial if they fulfill the inclusion and exclusion criteria of the trial. The inclusion and exclusion criteria are based upon those of the SCOT trial for adult dcSSc patients, which is the Phase 3 clinical trial in the United States comparing autologous HSCT to monthly high dose cyclophosphamide (CY) alone.

SUMMARY:
This phase I/II pilot trial seeks to demonstrate that prolonged administration of Campath-1H without prior marrow or stem cell harvesting can result in immunoablation similar to that achieved by hematopoietic stem cell transplantation (HSCT) from either bone marrow or peripheral blood stem cell sources in children and adolescents with severe treatment refractory systemic sclerosis (SSc).

DETAILED DESCRIPTION:
Patients, 8 to18 years of age, will be included if they have a proven diagnosis of diffuse cutaneous or systemic SSc as defined by the ACR criteria with evidence of active inflammatory disease Plus at least 1 of the following:SSc-related pulmonary disease with forced vital capacity (FVC) or hemoglobin-adjusted DLCO < 70% and evidence of alveolitis by high-resolution CT scan or bronchoalveolar lavage.

OR:History of SSc-related renal crisis or disease, not active at the time of screening

OR:Moderate to severe upper and/or lower gastrointestinal involvement

AND:Unacceptable toxicity or steroid dependence > 0.3 mg/kg/d,

OR:Failure to respond to, or unacceptable toxicity of MTX > 1mg/kg in combination with cyclosporine or azathioprine or cyclophosphamide 2 kg/d or Rituximab 375 mg/m2 x 4 doses or Imatinib 800 mg/

OR:Disease recurrence after tapering medication above

ELIGIBILITY:
4.2 Inclusion/Exclusion criteria 4.2.1 Inclusion criteria

* 8 to 21 years of age, inclusive
* Diffuse, cutaneous dcSSc as defined by the ACR criteria with evidence of active inflammatory disease.
* Plus at least 1 of the following:

  * dcSSc-related pulmonary disease with forced vital capacity (FVC) or hemoglobin-adjusted DLCO < 70% and evidence of alveolitis by high-resolution CT scan or bronchoalveolar lavage

OR

o History of SSc-related renal crisis or disease, not active at the time of screening

OR

* Moderate to severe upper and/or lower gastrointestinal involvement AND
* Unacceptable toxicity or steroid dependence > 0.3 mg/kg/d
* Failure to respond to, or unacceptable toxicity of MTX > 1mg/kg in combination with cyclosporine or azathioprine or cyclophosphamide or Rituximab 375 mg/m2 x 4 doses or Imatinib 800 mg/d or tocilizumab 8 mg/kg for at least 3 doses.
* Disease recurrence after tapering medication above (in #4)

4.2.2 Exclusion Criteria

* Pulmonary, cardiac, hepatic, or renal impairment that would limit therapy and compromise survival includes, but is not restricted to, any of the following:

  * Severe pulmonary dysfunction: hemoglobin-corrected DLCO < 45%, DLCO <4 mL/mmHg/min/L or pO2 < 70 mm Hg or pCO2, ≥ 45 mm Hg without supplemental O2 sat 92% at rest without supplemental O2
  * Significant pulmonary hypertension
  * Uncontrolled clinically significant arrhythmias
  * NYHA heart failure class IV
  * LVEF < 50% by echo or prior insertion of a pacemaker or cardioverter-defibrillator
  * End-stage renal disease (GFR<50 ml/min/1.73 m2 or creatinine . 2 mg/dl; estimated CrCl < 40 mL/min or active, untreated dcSSc renal crisis at time of enrollment
  * Active hepatitis (ALT, AST, or bilirubin > 2x ULN)
* Active gastric antral vascular ectasia (GAVE, "watermelon stomach")
* 2 mg/kg/day prednisone or equivalent within 30 days of treatment
* Unwilling or unable to discontinue DMARDs for treatment of dcSSc
* Co-morbid illnesses with an estimated median life expectancy < 5 Years
* Active uncontrolled infection
* Positive serology for hepatitis B or C, HIV
* ANC < 1500 cells/µL, platelets < 120,000 cells/µL, Hct < 27% or Hgb < 9.0 g/dL
* Malignancy within the previous 2 years, excluding treated skin cancer
* Myelodysplasia
* Uncontrolled hypertension
* History of hypersensitivity to murine or E. coli proteins
* Pregnancy or unwilling to use contraceptive methods for at least 15 months
* Steroid dependence: > 2mg/kg/day, prednisone or equivalent within 30 days prior to treatment
* History of substance abuse within the last 5 years
* History or presence of 2nd autoimmune disease requiring immunosuppressive therapy that has a substantial risk of recurrence
* Demonstrated lack of compliance with prior medical care
* Lack of rehabilitation potential

4.3 SSc patients, who fulfill the inclusion criteria, will then be assessed for residual thymic function since our previous study of pediatric dcSSc patients demonstrated that the dcSSc patients had decreased thymic function as compared to age matched controls as measured by the proportion of naïve CD4+ T lymphocytes (CD4+, CD31+), recent thymic emigrants (RTE). (5) Patients with less than 40% RTE will be excluded because of concerns about their ability to reconstitute their immune system after immune ablation.

4.4 dcSSc patients, who fulfill the screening criteria, will be consented for entry into the clinical trial.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients, 8 to18 years of age, will be included if they have a proven diagnosis of diffuse cutaneous or systemic SSc as defined by the ACR criteria with evidence of active inflammatory disease
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-04; Primary Completion 2018-08-02 (Actual); Study Completion 2018-09-02 (Actual)

PRIMARY OUTCOMES:
Primary outcome | 2 years
  To determine why the extended administration of Campath-1H results in immune ablation in some patients and immunosuppression in others, Number of Participants with Adverse Events as a Measure of Safety and Tolerability Campath-1H antibody levels during and after the completion of the Campath administration. (47) Thus, both the peak Campath-1H levels as well as the duration of circulating Campath will be determined.
Campath | The site will follow patients for 6 months post adverse event.
  Number of Participants with Adverse Events as a Measure of Safety and Tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Marzan, MD, Principal Investigator — Children's Hospital Los Angeles

IPD SHARING:
Plan to Share IPD: No